CLINICAL TRIAL: NCT03246984
Title: A Post Market Surveillance Multi-center Prospective Study to Evaluate the Safety and Efficacy of the VasQ External Support for Arteriovenous Fistula
Brief Title: VALUE- Vascular Access Laminate eUropean Experience. A Post Market Surveillance Study to Assess the Safety and Effectiveness of VasQ
Acronym: VALUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laminate Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD0097
Record Dates: First submitted 2017-08-03; First posted 2017-08-11 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Arterio-Venous Fistula; Kidney Failure, Chronic; Kidney Diseases; Renal Failure Chronic; ESRD; Arteriovenous Fistula Thrombosis
MeSH Terms: conditions — Arteriovenous Fistula; Kidney Failure, Chronic; Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VasQ device implantation (Experimental)
  Interventions: Device: VasQ

INTERVENTIONS:
Device: VasQ — VasQ device implantation in patients with a new brachiocephalic or radiocephalic fistula creation.

SUMMARY:
This is a prospective single arm study enrolling patients who are scheduled for creation of a new Brachiocephalic or Radiocephalic AV fistula. Up to 80 patients will be enrolled, 50 with upper arm AV fistula and 30 with forearm AV fistula. All patients will be implanted with the VasQ device, a subcutaneous arteriovenous conduit support for vascular access. The follow up period in this study will be for a duration of 12 months, with follow up visits scheduled at 1, 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred for creation of a new brachiocephalic or radiocephalic fistula who consent to take part in the study.
2. Age 18-80 years
3. Male and female participants
4. Patients willing and able to attend follow up visits over a period of 12 months

Exclusion Criteria:

1. Patients with the planned index procedure being a revision surgery of an existing fistula.
2. Target Brachial artery smaller than 2.5 mm or larger than 6 mm or Radial artery smaller than 2.5 mm or larger than 4 mm in outer diameter by preoperative ultrasound
3. Target vein outer diameter smaller than 2.5 mm by preoperative ultrasound
4. Significantly stenotic target vein on the side of surgery (≥50%) as diagnosed on pre-op ultrasound (scan should include the area between the planned anastomosis site and the Axillary vein)
5. Unusual anatomy or vessel dimensions (observed on pre-operative US or intraoperatively) and which preclude adequate fit of the VasQ.
6. Patients with prior central venous stenosis or obstruction on the side of surgery
7. Depth of vein greater than 8 mm (on ultrasound) on side of surgery
8. Known coagulation disorder
9. Congestive heart failure NYHA class ≥ 3
10. Prior steal on the side of surgery as evident from the patient's medical history
11. Known allergy to nitinol
12. Life expectancy less than 18 months
13. Patients expected to undergo kidney transplant within 6 months of enrollment
14. Women of child bearing potential without documented current negative pregnancy test
15. Inability to give consent and/or comply with the study follow up schedule

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Primary patency of AV fistula | 6 months post AVF creation
  Freedom from any intervention designed to maintain or reestablish patency since device placement and demonstrate flow on Doppler US.
  1 = Success = Intervention free access patency determined by Doppler ultrasound.
  0 = Failure = Access occluded determined by Doppler ultrasound and/or underwent intervention

CONTACTS AND LOCATIONS:
Overall Officials: Noam Zilberman, Study Director — Laminate Medical Technologies Ltd.
Locations (11):
- Institut Mutualiste Montsouris, Paris, France
- Germany (8):
  - Universitätsklinikum Augsburg, Augsburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Königin Elisabeth Krankenhaus Herzberge, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - University Hospital Cologne, Cologne
  - Universitaetsklinikum Jena, Jena
  - Klinikum Ernst von Bergmann gemeinnützige GmbH, Potsdam
  - Harzklinikum Dorothea Christiane Erxleben, Wernigerode
- Hospital Clinic of Barcelona, Barcelona, Spain
- Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chemla E, Velazquez CC, D'Abate F, Ramachandran V, Maytham G. Arteriovenous fistula construction with the VasQ external support device: a pilot study. J Vasc Access. 2016 May 7;17(3):243-8. doi: 10.5301/jva.5000527. Epub 2016 Apr 14. PMID 27079670
- See also: Related Info — http://www.laminatemedical.com/